CLINICAL TRIAL: NCT05995691
Title: A Randomized, Single-blind, Single-dose, 2-Arm, Parallel-group Study to Determine the Pharmacokinetic Bioequivalence of ABP 501 and Adalimumab (Humira®) in Healthy Adult Japanese Subjects
Brief Title: Study to Determine the Pharmacokinetic (PK) Bioequivalence of ABP 501 and Adalimumab (Humira®) in Healthy Adult Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20120176
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: ABP 501; Adalimumab; Humira®
MeSH Terms: interventions — ABP 501; Adalimumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABP 501 (Experimental): Participants will receive a single dose of ABP 501
  Interventions: Drug: ABP 501
- Adalimumab (Active Comparator): Participants will receive a single dose of adalimumab
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: ABP 501 — SC injection
  Arms: ABP 501
Drug: Adalimumab — SC injection
  Other Names: Humira®
  Arms: Adalimumab

SUMMARY:
The primary objective of this study is to determine the bioequivalence of ABP 501 (subcutaneous [SC] injection) compared to adalimumab (SC injection) as assessed principally by the area under the serum concentration-time curve from time 0 extrapolated to infinity (AUCinf), and maximum observed serum concentration (Cmax) in Japanese participants.

ELIGIBILITY:
Inclusion Criteria

1. Participants must sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved ICF before any study-specific procedures are performed.
2. Healthy adult male and female Japanese participants between 18 and 45 years of age, inclusive, at the time of screening.
3. Body mass index (BMI) between 16.0 and 25.0 kg/m2, inclusive, at screening and Day -1.
4. Normal or clinically acceptable physical examination, clinical laboratory test values, vital signs, and electrocardiogram (ECG) (12-lead ECG reporting heart rate and RR, PR, QRS, QT, and QTc intervals), as determined by the investigator, at screening. Physical examination, vital signs, body weight and BMI, clinical laboratory tests, pregnancy test, urinalysis, urine drug screen, and alcohol screen will be repeated on Day -1 (see Table 2-1) and must also be normal or clinically acceptable, as deemed by the investigator.
5. Participants must be current on immunizations per local standards.
6. Participants must be first- or second-generation Japanese:

   * First-generation Japanese are participants who may be living outside of Japan but were born in Japan to parents of Japanese descent
   * Second-generation Japanese are participants who were born outside of Japan to first-generation Japanese parents

Exclusion Criteria

1. Women of childbearing potential who are unwilling to practice a highly effective method of birth control for the duration of the study and for 5 months following treatment with the investigational product or until the scheduled end-of-study (EOS) (whichever is longer). Acceptable methods of effective birth control include:

   * Abstinence
   * Surgical methods: bilateral tubal ligation or vasectomy for the male sexual partner
   * Hormonal methods
   * Intrauterine device (IUD)
   * Two barrier methods (one by each partner)

     * The male must use a condom (latex or other synthetic material)
     * The female may select one of the following barrier methods: diaphragm, cervical, or contraceptive sponge
2. Women who are lactating or breastfeeding.
3. Women with a positive pregnancy test.
4. Women planning to become pregnant during the study or within 5 months following treatment with investigational product.
5. History or evidence of a clinically significant disorder (including psychiatric), condition, or disease that, in the opinion of the investigator, would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
6. History or evidence of any bacterial, viral, parasitic, or systemic fungal infections within the past 30 days prior to investigational product administration (eg, upper respiratory tract infection, viral syndrome, flu-like symptoms). Exception: a simple, short-duration common cold within the past 14 days prior to investigational product administration.
7. A recent infection (within 6 months of randomization) requiring inpatient hospitalization or intravenous antibiotics.
8. Known positive tuberculin skin test or exposure to an individual with tuberculosis (TB) or positive QuantiFERON® test or local equivalent (eg, T-Spot®) consistent with previous exposure to TB prior to or during screening (if not treated with appropriate chemoprophylaxis).
9. Tuberculosis or fungal infection seen on available chest x-ray taken within 6 months of screening or at screening.
10. History of malignancy of any type, other than surgically excised nonmelanomatous skin cancers, within 5 years prior to randomization.
11. Positive test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at screening.
12. Positive screen for alcohol and/or potential drugs of abuse at screening or prior to randomization.
13. Receiving or has received any investigational drug (or is currently using an investigational device) within 30 days or 5 half-lives (whichever is longer), prior to receiving investigational product.
14. Use of any over-the-counter (OTC) or prescription medications within the 14 days or 5 half-lives (whichever is longer), prior to receiving investigational product. Acetaminophen (up to 2 g per day and not more than 4 g per week) for analgesia will be allowed. Hormonal contraceptives are allowed.
15. All herbal medicines (eg, St. John's wort) and supplements consumed by the participant within the 30 days prior to receiving investigational product, and continuing use if applicable, will be reviewed by the investigator and the ICON medical monitor. Written documentation of this review and Amgen acknowledgment of the decision made with respect to eligibility is required for participant participation.
16. Donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months of screening.
17. Received live vaccines ≤ 3 months prior to investigational product administration or are scheduled to receive a live vaccine within 3 months following treatment with investigational product.
18. Known or suspected sensitivity to products derived from mammalian cell lines.
19. Known allergy to natural rubber (latex).
20. Previously received adalimumab or a biosimilar of adalimumab.
21. History of alcohol and/or substance abuse within the last 12 months from screening.
22. Participants who use > 10 cigarettes per day within the last 3 months or not able to abide by the smoking policy of the clinical pharmacology unit (CPU).
23. Inability or unwillingness to reside at the CPU for 2 consecutive days or inability to be available for follow-up assessments or protocol-required procedures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2015-12-04 (Actual); Study Completion 2015-12-04 (Actual)

PRIMARY OUTCOMES:
AUCinf of ABP 501 | Day 1 to Day 63
Cmax of ABP 501 | Day 1 to Day 63
AUCinf of Adalimumab | Day 1 to Day 63
Cmax of Adalimumab | Day 1 to Day 63

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Day 1 to Day 63
  Any clinically significant changes in vital signs or clinical laboratory test results after the dose of treatment will be recorded as TEAEs.
Number of Participants With Anti-drug Antibodies (ADA) | Day 1 to Day 63
Terminal Phase Elimination Half-life (t1/2) of ABP 501 | Day 1 to Day 63
t1/2 of Adalimumab | Day 1 to Day 63
Time at Which the Maximum Observed Serum Concentration is Observed (Tmax) of ABP 501 | Day 1 to Day 63
Tmax of Adalimumab | Day 1 to Day 63
Area Under the Serum Concentration-time Curve from Time 0 to the Last Quantifiable Concentration (AUClast) of ABP 501 | Day 1 to Day 63
AUClast of Adalimumab | Day 1 to Day 63

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com